CLINICAL TRIAL: NCT01470534
Title: Investigating Whether the Magnitude of Postoperative Inflammatory and Insulin Resistant Responses is Related to Body Composition and Physiological Function of Skeletal Muscle & Adipose Tissue
Brief Title: Mechanisms Underlying Postoperative Insulin Resistance and Inflammation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11040
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Obesity
Keywords: Dietary supplement; Carbohydrate loading; Insulin resistance; Surgery
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal body weight (Experimental)
  Interventions: Dietary Supplement: carbohydrate drink; Procedure: Muscle biopsy; Procedure: Blood sampling
- Obese (Experimental)
  Interventions: Dietary Supplement: carbohydrate drink; Procedure: Muscle biopsy; Procedure: Blood sampling
- Normal Body Weight placebo (Placebo Comparator): Participants of mormal body weight given placebo
  Interventions: Procedure: Muscle biopsy; Procedure: Blood sampling; Dietary Supplement: Placebo
- Obese placebo (Placebo Comparator): Participants who are obese given placebo
  Interventions: Procedure: Muscle biopsy; Procedure: Blood sampling; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: carbohydrate drink — carbohydrate drink
  Arms: Normal body weight; Obese
Procedure: Muscle biopsy — Open muscle biopsy
Procedure: Blood sampling — Venopuncture
Dietary Supplement: Placebo
  Arms: Normal Body Weight placebo; Obese placebo

SUMMARY:
Having an operation places an enormous burden on the body, leading to the development of inflammation and so called 'insulin resistance'. Insulin resistance means the body is unable to respond to important hormones that control use of energy. Recent studies have shown that patients who develop 'higher' insulin resistance and inflammation have more serious complications and take longer to recover after surgery. The investigators do not know what controls the development of insulin resistance and inflammation after surgery. Similarly, the investigators do not know why certain patients develop much more insulin resistance and inflammation than others, even though they have the same operation.

The main purpose of the study is to try to find out which patients are prone to developing greater 'amounts' of insulin resistance and inflammation. The investigators also want to find out whether the investigators can reduce the 'amount' of insulin resistance and inflammation in these patients (for example by giving them carbohydrate [sugar-based] drinks before surgery - these have been shown to reduce insulin resistance in some patient groups).

Information from this study should improve the way the investigators prepare patients before surgery and this should help to improve patient outcomes following surgery (by reducing complications and speeding recovery after major surgery).

DETAILED DESCRIPTION:
Interested participants who are undergoing abdominal (tummy) surgery will be recruited from surgical clinics. They will be asked to attend the Greenfield Human Physiology Laboratory where they will be asked to complete two questionnaires. In addition, a sample of blood, and a small sample of muscle and fat from their thigh will be taken. They will undergo a low dose X-ray (DXA scan) and an insulin clamp. The insulin clamp involves being connected to an insulin and glucose drip for around four hours during which their blood pressure and pulse is monitored and regular blood samples are taken.

Participants will be allocated randomly to one of two groups. One group will receive a carbohydrate (sugar) drink before surgery and the other group will receive a dummy (placebo) drink.

On the day of surgery, pre-operative checks and assessment will proceed as normal. After the participant is asleep under anaesthetic, a blood sample and tummy muscle and fat samples will be taken by the surgeon through the surgical incision. At the end of surgery, another blood sample and muscle and fat samples from the tummy and thigh will be taken while the participant is still under anaesthetic.

On the day after surgery, a further blood test and tummy and thigh muscle and fat sample will be taken. Participants will also undergo another insulin clamp.

The research team will follow participants' progress after surgery, but the decision to allow them home will be made by the medical team responsible for their care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 yrs
* Correct BMI and waist circumference criteria : Obese group - BMI ≥30 AND waist circumference ≥94 cm in men and ≥ 80 cm in women, Non obese group - BMI 18.5-25 AND waist circumference ≤94cm in men and ≤80 cm in women Due to undergo elective major abdominal surgery ASA I-III Caucasian patients Able to give informed consent and comply with study protocol

Exclusion Criteria:

* History of significant preoperative weight loss (>10% over preceding 3 weeks)

  * Clinical history of pulmonary aspiration
  * Known gastro-oesophageal reflux disease (GORD) or hiatus hernia
  * History of difficult intubation or conditions leading to the latter such as: previous neck radiotherapy/rheumatoid arthritis/presence of thyroid goitre
  * Metabolic disorders (e.g. diabetes mellitus, thyroid disease, Cushing's Syndrome)
  * Simultaneous participation in another clinical study or involvement in a clinical study within the preceding 3 months,
  * Patients with suspicion of alcohol/drug abuse
  * Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Within subject differences in perioperative insulin sensitivity (M-value, corrected for insulin concentrations) amongst obese, non-obese, carbohydrate loaded and non-carbohydrate loaded patients. | 2 weeks

SECONDARY OUTCOMES:
Correlation between body composition and changes in perioperative insulin sensitivity | 2 weeks
Differences in inflammatory cytokine gene expression | 2 months
Differences in muscle and fat genes and proteins controlling carbohydrate/fat oxidation and insulin signalling | 3 months
Differences activities of muscle and fat enzymes involved in carbohydrate/fat/carnitine metabolism | 2 months
Differences in the aforementioned between peripheral and central fat and muscle | 2 months
The incidence of post-operative infectious and non-infectious complications | 30 days
Length of hospital stay (difference between groups) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom